CLINICAL TRIAL: NCT00661323
Title: Left Ventricular Strain Quantification From 4D Echocardiography
Brief Title: Evaluating a New Echocardiography Imaging Procedure for Evaluating Heart Function
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0608001734_B; R01HL082640 (NIH)
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2016-06

CONDITIONS: Ischemia; Myocardial Infarction; Ischemic Heart Disease
MeSH Terms: conditions — Ischemia; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Healthy volunteers will be recruited through the use of an approved study recruitment flyer.
- 2: Chemotherapy patients will be approached at the time of their nuclear scan to rule out cardiac disease prior to chemotherapy. These patients will be referred to the study by their doctor for the assessment of heart function.

SUMMARY:
Magnetic resonance imaging (MRI) and echocardiography are two imaging methods that are used to obtain pictures of the heart and assess heart function. This study will evaluate a new, four-dimensional echocardiography approach of obtaining heart images to determine if it is as effective at evaluating heart function as MRI.

DETAILED DESCRIPTION:
MRI is a non-invasive method of obtaining images of the body. An MRI is conducted by having a person lie down on a narrow table, which then slides into a large tunnel-like tube. Powerful magnets and radio waves scan the body and a computer records the resulting signals. An echocardiography is a non-invasive ultrasound test that uses sound waves to create images of the heart. It is performed by having a doctor move a wand-like device over a patient's chest. The device then converts sound waves into pictures of the heart. Currently, a special MRI technique is used to evaluate heart function; however, MRI is expensive and cannot be used on critically ill patients. Echocardiography can be performed at a patient's bedside and it may be a more effective way of assessing heart function. The purpose of this study is to determine the effectiveness of a new four-dimensional echocardiography approach at evaluating heart function. Results from this study may be used to diagnose and treat patients more effectively in the future.

This study will enroll healthy people who do not have heart disease and people who are receiving chemotherapy who do not have heart disease. Participants will have a physical examination and a medical records review. MRI scans and a four-dimensional echocardiography of the heart will be performed. There will be no additional study visits.

ELIGIBILITY:
Inclusion Criteria:

* No evidence of underlying cardiac disease based on history or electrocardiogram (ECG)
* Adequate intravenous access in one arm

Exclusion Criteria:

* Pregnant or breastfeeding; if pre-menopausal, not practicing acceptable method of birth control
* History of any other medical condition that is likely to hinder study conduct or pose a safety concern, in the opinion of the investigator
* History of cardiac disease, including heart attack or heart valve disease
* Uncontrolled high blood pressure, defined as systolic blood pressure higher than 160 mm Hg and/or diastolic pressure higher than 100 mm Hg
* Abnormal ECG or chest pain syndrome
* Claustrophobia
* Resting heart rate greater than 110 bpm
* Unable to undergo MRI procedure (e.g., pacemaker, metallic implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will consist of two groups:
  1. Normal volunteers will be recruited through the use of an approved study recruitment flyer.
  2. Chemotherapy patients will be approached at the time of their nuclear scan to rule out cardiac disease prior to chemotherapy. These patients will be referred to the study by their doctor for the assessment of heart function.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Establish baseline strain patterns for future studies evaluating alterations in left ventricular strain/strain rates associated with regional myocardial ischemia and injury | Measured at participants' study visit

CONTACTS AND LOCATIONS:
Overall Officials: Albert J. Sinusas, MD, Principal Investigator — Yale University
Locations (1):
- Yale University/Magnetic Resonance Research Center (MR-TAC)/Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Constable RT, Rath KM, Sinusas AJ, Gore JC. Development and evaluation of tracking algorithms for cardiac wall motion analysis using phase velocity MR imaging. Magn Reson Med. 1994 Jul;32(1):33-42. doi: 10.1002/mrm.1910320106. PMID 8084235
- [Background] Duncan J, Shi P, Constable T, Sinusas A. Physical and geometrical modeling for image-based recovery of left ventricular deformation. Prog Biophys Mol Biol. 1998;69(2-3):333-51. doi: 10.1016/s0079-6107(98)00014-5. PMID 9785945
- [Background] Shi P, Sinusas AJ, Constable RT, Ritman E, Duncan JS. Point-tracked quantitative analysis of left ventricular surface motion from 3-D image sequences. IEEE Trans Med Imaging. 2000 Jan;19(1):36-50. doi: 10.1109/42.832958. PMID 10782617
- [Background] Papademetris X, Sinusas AJ, Dione DP, Duncan JS. Estimation of 3D left ventricular deformation from echocardiography. Med Image Anal. 2001 Mar;5(1):17-28. doi: 10.1016/s1361-8415(00)00022-0. PMID 11231174
- [Background] Sinusas AJ, Papademetris X, Constable RT, Dione DP, Slade MD, Shi P, Duncan JS. Quantification of 3-D regional myocardial deformation: shape-based analysis of magnetic resonance images. Am J Physiol Heart Circ Physiol. 2001 Aug;281(2):H698-714. doi: 10.1152/ajpheart.2001.281.2.H698. PMID 11454574
- [Background] Meyer FG, Constable RT, Sinusas AJ, Duncan JS. Tracking myocardial deformation using phase contrast MR velocity fields: a stochastic approach. IEEE Trans Med Imaging. 1996;15(4):453-65. doi: 10.1109/42.511749. PMID 18215927
- [Background] Shi P, Sinusas AJ, Constable RT, Duncan JS. Volumetric deformation analysis using mechanics-based data fusion: Applications in cardiac motion recovery. International J Computer Vision 35:87-107, 1999